CLINICAL TRIAL: NCT00526682
Title: The Effect of Combining Cissus Quadrangularis and Irvingia Gabonensis on Obesity and Obesity Related Diseases
Brief Title: The Use of Irvingia Gabonensis (Bush Mango)and Cissus Quadrangularis to Reduce Weight and Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gateway Health Alliance (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GHACT010
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Obesity; Overweight; Dyslipidemia
Keywords: Antiobesity; Weight loss
MeSH Terms: conditions — Obesity; Overweight; Dyslipidemias; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Comparison of actives for synergy
  Interventions: Dietary Supplement: Irvingia/cissus combo

INTERVENTIONS:
Dietary Supplement: Irvingia/cissus combo
  Other Names: Irvingia cissus combo

SUMMARY:
Hypothesis: Cissus quadrangularis as well as Irvingia gabonensis are used in weight management and related conditions. This study set out to investigate if a combination of the two could have additional benefits to overweight and obese people.

DETAILED DESCRIPTION:
To assess and compare the effects of administration of Cissus quadrangularis (Linn) and a Cissus quadrangularis /Irvingia gabonensis combination on body weight blood pressure, fasting blood glucose, plasma total and LDL cholesterol in 72 overweight and obese subjects.

The study was a 10 week randomized, double-blind, placebo-controlled design, involving 72 obese or overweight participants. Participants were randomly divided into three groups (24 participants/ group):

Group 1 - Placebo; Group 2 - Cissus quadrangularis (CQ); Group 3 - Cissus quadrangularis and Irvingia gabonensis (CQ-IG).

The placebo (250mg) or active formulations ((150 mg CQ and 250 mg CQ-IG) were administered twice daily before meals. Weight as well as fasting blood was taken at baseline, and at 4, 8 and 10 weeks.

No major dietary changes or exercises were suggested during the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI>26kg/m2

Exclusion Criteria:

* Diabetics
* Pregnant and lactating
* Subjects on any other weight loss program
* Following any specific low calorie diet

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Weight change | 10 weeks

SECONDARY OUTCOMES:
Blood lipids Body fat Fasting blood glucose | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julius E OBEN, PhD, Principal Investigator — University of Yaounde 1